CLINICAL TRIAL: NCT06968702
Title: Project ICOPE Brazil: Assessment of Intrinsic Capacity in Older Adults as a Basis for Implementation of the WHO ICOPE Strategy in the Unified Health System.
Brief Title: Project ICOPE Brazil: Assessment of Intrinsic Capacity in Brazilian Older Adults
Acronym: ICOPE-BR
Status: Not yet recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Ferriolli, Full Professor, University of Sao Paulo
Other Study IDs: EFerriolli
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Intrinsic Capacity; Frailty; Aging; Healthy Aging; Functional Ability; Mobility and Independence; Cognitive Ability, General; Cognitive Impairment; Sensory Hearing Loss; Sensory Deficits; Visual Acuity; Visual Impairment; Mood Disorders; Depressive Symptoms; Vitality; Nutritional Risk; Nutrition Assessment
Keywords: Instrinsic Capacity; Functional Ability; ICOPE; Aging trends; Older Adults; Frailty; Cognitive Impairment; Mobility; Sensory; Vitality; Psychological; Cohort; healthy aging; public health
MeSH Terms: conditions — Frailty; Cognitive Dysfunction; Hearing Loss, Sensorineural; Vision Disorders; Mood Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Plasma specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community-dwelling older adults: Population Community-dwelling people aged ≥ 60 years registered in the participating primary health care units, and domiciled in their respective coverage area. Participants do not have to be active patients to be invited.
  We will create a random order from the lists of users registered in each health care unit involved in the project to invite participants. This approach ensures a systematic random sampling strategy to avoid participants' enrollment by convenience and its related selection bias.
  Participants will be invited via telephone or home visits, following the order established by the randomization list, until we reach the minimum expected number of participants for each center. For centers that need to enroll participants from two or more health care units to achieve the minimum expected sample size of 202 participants, it is necessary to consolidate the user lists from these units into a single list before randomization.

SUMMARY:
The ICOPE Brazil study aims to understand aging trajectories in Brazil, especially healthy aging trends based on intrinsic capacity, a collective of mental and physical capacities one may have to maintain their functional ability to execute daily life activities. Tests and questionnaires will be applied to collect data on mobility capacity, cognitive capacity, nutritional status, vision, and hearing (sensorial) capacities, and mental health. These assessments are in consonance with what the World Health Organization proposed in the Integrated Care for Older People Program (ICOPE). Participants will be followed up for three years, and the primary outcomes of interest are loss of intrinsic capacity, mobility impairment, cognitive impairment, incident depressive symptoms, loss of functional ability, incident frailty, incident sarcopenia, incident falls, hospitalization, multimorbidity, and mortality.

DETAILED DESCRIPTION:
The ICOPE Brazil study is a prospective, longitudinal cohort study designed to investigate the trajectories of aging among older adults in Brazil, with a particular emphasis on healthy aging as defined by the World Health Organization (WHO). The central conceptual framework guiding this study is "intrinsic capacity," a multidimensional construct encompassing an individual's physical and mental capacities that contribute to the maintenance of functional ability in later life.

Data collection will involve the administration of standardized tests and structured questionnaires to assess five core domains of intrinsic capacity: mobility, cognitive function, nutritional status, sensory capacities (vision and hearing), and psychological well-being. These domains reflect the recommendations outlined in the WHO's Integrated Care for Older People (ICOPE) program, which aims to promote healthy aging and support the functional ability of older populations globally.

Participants will be followed for a total duration of three years, with periodic assessments to monitor changes over time. The primary outcomes of interest include: decline in intrinsic capacity, mobility impairment, cognitive impairment, onset of depressive symptoms, loss of functional ability, incident frailty, incident sarcopenia, incidence of falls, hospitalizations, multimorbidity, and all-cause mortality. Data generated from this study will inform public health strategies, clinical guidelines, and policy development for aging populations in Brazil and other similar settings.

ELIGIBILITY:
Inclusion Criteria:

* People aged ≥ 60 years, with no age limit;
* Being registered (with available contact information) in the participating health care units;
* Being available to go in person to the data collection sites for the assessments.

Exclusion criteria

* Inability to access the data collection site;
* Severe neurologic and/or cognitive impairments that preclude interaction with the evaluators to complete the proposed tests and data collections;
* Advanced serious illness or under palliative care:

Clinical Frailty Scale (CFS)20 score of 8 (severely frail) or 9 (terminally ill).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling people aged ≥ 60 years who are users of the public health system, and registered in the participating primary health care units domiciled in their respective coverage area.
Sampling Method: Non-Probability Sample
Enrollment: 3838 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Loss of Intrinsic Capacity | Participants will be reassessed by a telehealth visit at 6, 18, 30 months using the ICOPE basic assessment strategy. In-person visits at 12, 24 and 36 months of follow up.
  Changes from baseline in Intrinsic Capacity domains over time. Mobility: delta of the Short Physical Performance Battery and its criterion. Cognition: delta of the Montreal Cognitive Assessment Score Vision: changes in visual acuity category assessed by the Snellen visual chart Hearing: changes in the Hearing Handicap Inventory For The Elderly category Nutrition/Vitality: changes in the Mini-nutritional risk category and the delta of its scores.
  Depressive Symptoms: changes in the Geriatric Depression Scale results.

SECONDARY OUTCOMES:
Major Geriatric Outcomes | Telehealth monitoring at 6, 18, 30 months of follow up. In-person visits at 12, 24, 36 months of follow up
  Major Geriatric Outcomes are:
  Loss of Functional Ability Incident Falls Incident Fractures Urinary Incontinence Incident Frailty Incident Sarcopenia Incident Dementia Moving to a long-term care or Nursing Home facility Hospitalization ED visits Death

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ferriolli, MD, MSc, PhD, Study Chair — University of Sao Paulo; Renato Bandeira de Mello, MD, MPH, PhD, Study Director — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Assessment of intrinsic capacity in the Brazilian older population and the psychometric properties of the WHO/ ICOPE screening tool: a multicenter cohort study protocol. Geriatr Gerontol Aging. 2024; https://doi.org/10.53886/gga.e0000166_EN
- See also: Study website — https://icopebrasil.org/
- See also: Study Protocol — https://cdn.publisher.gn1.link/ggaging.com/pdf/en_v18e000166.pdf